CLINICAL TRIAL: NCT05001360
Title: Evaluating the Efficacy and Safety of FMT Capsules XBI-302 Combined With Nivolumab in the Treatment of Anti-PD-1/L1 Resistant Gastric Cancer
Brief Title: Study of FMT Combined With Nivolumab in Gastric Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not get the IRB approval.
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-022
Record Dates: First submitted 2021-07-26; First posted 2021-08-11 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-07

CONDITIONS: Gastric Adenocarcinoma; Esophagogastric Junction Adenocarcinoma; Esophagus Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Nivolumab; Fecal Microbiota Transplantation; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XBI-302 + Nivolumab (Experimental): FMT capsules XBI-302 will be administered orally every two weeks for 12 weeks and then every four weeks for 12 weeks. Nivolumab will be intravenously infused every two weeks for 24 weeks.
  Interventions: Drug: XBI-302 + Nivolumab

INTERVENTIONS:
Drug: XBI-302 + Nivolumab — After gut preparation, a single dose of FMT will be performed via oral administration. Subsequently, nine combined treatment cycles that composed of anti-PD-1 infusions (Nivolumab at 240 mg, q2w) and additional FMT capsules, and 3 single treatment cycles of anti-PD-1 infusions will be administered.
  Other Names: FMT + PD-1 inhibitor

SUMMARY:
This study is a single-arm, single center study. The purpose of this study is to evaluate the efficacy and safety of FMT capsules XBI-302 combined with Nivolumab in the treatment of anti-PD-1/L1 resistant gastric cancer.

DETAILED DESCRIPTION:
The primary purpose of this single-arm, open-label, single center trial is to evaluate the efficacy and safety of XBI-302 combined with Nivolumab in the treatment of anti-PD-1/L1 resistant gastric cancer.

During treatment period, all eligible subjects will receive XBI-302 with Nivolumab following gut preparation. The imaging evaluation of efficacy will be performed every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study and provide written informed consent
* Age ≥ 18 years and ≤70 years, male or female
* Pathological confirmed locally advanced, unresectable or metastatic gastric adenocarcinoma, esophagogastric junction adenocarcinoma and lower esophagus adenocarcinoma that are resistant to anti-PD-1/L1 antibodies
* Able and willing to provide tumor tissue
* At least one measurable extracranial target lesion according to iRECIST
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥3 months

Exclusion Criteria:

* History of other primary malignancies within 5 years except adequately treated in situ carcinoma of the cervix or non-melanoma carcinoma of the skin
* Had systemic diseases that were difficult to control within 4 weeks prior to screening
* History of anti-PD-1 antibodies related adverse reactions that led to the permanent withdrawal of anti-PD-1 therapy
* History of coagulation disorders
* Mechanical or paralytic obstruction of the gastrointestinal tract
* Anticipated to receive a great number of antibiotics during study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 24 weeks
  iCR + iPR + iSD rate according to iRECIST criteria

SECONDARY OUTCOMES:
Disease control rate | 6, 12, 18 weeks
  iCR + iPR + iSD rate according to iRECIST criteria
Objective response rate | 24 weeks
  iCR + iPR rate according to iRECIST criteria
Changes of intestinal microbiota characteristics between responders and non-responders | 24 weeks
  To compare the change of intestinal microbiota characteristics between responders and non-responders
Changes of related immune cells in peripheral blood between responders and non-responders | 12 weeks
  To compare the change of related immune cells in peripheral blood between responders and non-responders
Change of CD8+T cell counts in tumor tissue between responders and non-responders | 6 weeks
  To compare the change of CD8+T cell counts in tumor tissue between responders and non-responders
Change of CD8+T cell counts in intestinal tissue between responders and non-responders | 6 weeks
  To compare the change of CD8+T cell counts in intestinal tissue between responders and non-responders
Incidence and severity of AEs that related to XBI-302 | 24 weeks
  Rate of adverse events and their severity that are determined to be related to XBI-302
Incidence and severity of immune related AEs | 24 weeks
  Rate and severity of irAEs

OTHER OUTCOMES:
OS | up to 2 years
  Overall survival defined as the time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No